CLINICAL TRIAL: NCT01496495
Title: A Study of ARRY-614 in Patients With Low or Intermediate-1 Risk Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-614-112
Record Dates: First submitted 2011-11-28; First posted 2011-12-21 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — pexmetinib

ARMS (1):
- ARRY-614 (Experimental)
  Interventions: Drug: ARRY-614, p38/Tie2 inhibitor; oral

INTERVENTIONS:
Drug: ARRY-614, p38/Tie2 inhibitor; oral — Part 1: multiple dose, escalating; Part 2: multiple dose, single schedule

SUMMARY:
This is a Phase 1 study during which patients with low or intermediate-1 risk myelodysplastic syndromes (MDS) will receive investigational study drug ARRY-614.

This study has 2 parts. In the first part, patients will receive increasing doses of study drug in order to achieve the highest dose of the study drug possible that will not cause unacceptable side effects. Approximately 50 patients from the US will be enrolled in Part 1 (Completed).

In the second part of the study, patients will receive the best dose of study drug determined from the first part of the study and will be followed to see what side effects and effectiveness the study drug has, if any, in treating the cancer. Approximately 30 patients from the US will be enrolled in Part 2 (Completed).

ELIGIBILITY:
Key Inclusion Criteria (Part 1 and Part 2):

* Diagnosis of MDS by bone marrow biopsy.
* International Prognostic Scoring System (IPSS) score of low or intermediate-1 risk MDS.
* May have received prior therapy for MDS.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1 or 2.
* Adequate liver and renal function.
* Additional criteria exist.

Key Exclusion Criteria (Part 1 and Part 2):

* History of bone marrow transplant.
* Treatment for MDS other than transfusions or a stable dose (≥ 4 weeks) of hematopoietic growth factors on the day of the first dose of study drug.
* Concomitant malignancies or previous malignancies with less than a 2-year disease-free interval at the time of enrollment.
* Treatment with an investigational medicinal product that is not expected to be cleared by the first dose of study drug or that has demonstrated to have prolonged side effects.
* Treatment with azacitidine or decitabine within 2 weeks prior to first dose of study drug.
* Chronic use (> 2 weeks) of greater than physiologic doses of corticosteroids (dose equivalent to > 20 mg/day of prednisone) within 4 weeks prior to first dose of study drug.
* Treatment with an immunomodulatory agent within 4 weeks prior to the first dose of study drug.
* Additional criteria exist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-03-18 (Actual)

PRIMARY OUTCOMES:
Establish the maximum tolerated dose (MTD) of study drug. | Part 1, 9 months
Characterize the safety profile of the study drug in terms of adverse events, clinical laboratory tests and electrocardiograms. | Part 1, 9 months; Part 2, 9 months
Characterize the pharmacokinetics (PK) of the study drug and a metabolite in terms of plasma concentrations. | Part 1, 9 months; Part 2, 9 months

SECONDARY OUTCOMES:
Assess the efficacy of the study drug in terms of response, time to response, duration of response, overall survival, hematologic improvement and platelet transfusion independence/reduction. | Part 1, 9 months; Part 2, 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Winship Cancer Institute, Atlanta, Georgia
  - Cleveland Clinic, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Su H, Jiang M, Senevirathne C, Aluri S, Zhang T, Guo H, Xavier-Ferrucio J, Jin S, Tran NT, Liu SM, Sun CW, Zhu Y, Zhao Q, Chen Y, Cable L, Shen Y, Liu J, Qu CK, Han X, Klug CA, Bhatia R, Chen Y, Nimer SD, Zheng YG, Iancu-Rubin C, Jin J, Deng H, Krause DS, Xiang J, Verma A, Luo M, Zhao X. Methylation of dual-specificity phosphatase 4 controls cell differentiation. Cell Rep. 2021 Jul 27;36(4):109421. doi: 10.1016/j.celrep.2021.109421. PMID 34320342